CLINICAL TRIAL: NCT05263687
Title: Cardio Pulmonary Exercise Testing (CPET) in Diseases and Health
Brief Title: Exercise Testing in Diseases and Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Principal Investigator, Gur Mainzer, Head of the pediatric cardiology department, The Baruch Padeh Medical Center, Poriya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0033-17-POR
Record Dates: First submitted 2022-02-13; First posted 2022-03-02 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Test (Experimental): maximal and anaerobic threshold cardiopulmonary parameters
  Interventions: Diagnostic Test: Maximal exercise test

INTERVENTIONS:
Diagnostic Test: Maximal exercise test — Each participants will conduct a spirometry test and exercise test on treadmill (using Modified Bruce Protocol) or cycle ergometer. Quark CPET metabolic cart (Cosmed, Rome, Italy) will be used to collect and analysis gas exchange, ECG, gas volume in addition rating of perceived exertion will be asked.

SUMMARY:
Cardiopulmonary exercise test (CPET) is a helpful tool for evaluation of aerobic exercise capacity and tolerance for variety of population. CPET provides a full assessment of the physiologic responses of the pulmonary, cardiovascular, muscular, and cellular oxidative systems to exercise. The test progression include a incremental stepwise (on treadmill) or ramp control protocol (on bike ergometer ) to exhaustion. Measurement of respiratory gas exchange i.e. oxygen uptake, carbon dioxide, minute ventilation, other variables while monitoring ECG, blood pressure, pulse oximetry and exertion perceived (Borg Scale) during an incremental test .

Aim: To compere exercise responses for maximal exercise testing with different population.

DETAILED DESCRIPTION:
Each participants will conducted an exercise test on treadmill using Modified Bruce Protocol) or cycle ergometer. Quark CPET metabolic cart (Cosmed, Rome, Italy) will be use to collect and analysis gas exchange. 10 minute after the graded exercise test Supra maximal exercise test (SMT) will be done for 2 minutes one stage (treadmill protocol) or 10% at cycle protocol higher than highest load achieved in the incremental test.

all outcome measurement will be collected. Exercise tolerance and responses will be assess using the data of : pulmonary gas exchange; cardiovascular performance, and skeletal muscle metabolism.

ELIGIBILITY:
Inclusion Criteria:

*Patient who invited to the clinic to do incremental maximal exercise test or healthy *Participants with no known significant health problems.

Exclusion Criteria:

* Acute fever
* Acute myocardial infarction within 2 to 3 days.
* Unstable angina not previously stabilized by medical therapy.
* Uncontrolled cardiac arrhythmias causing symptoms or hemodynamic compromise.
* Symptomatic severe aortic stenosis.
* Uncontrolled symptomatic heart failure.
* Inability to perform exercise Orthopedic impairment severely compromising exercise performance.

Ages: 4 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2017-08-30 (Actual); Primary Completion 2025-03-19 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximal Oxygen consumption | through study completion, an average of 1 year
  the maximum amount of oxygen that an individual can utilize during intense or maximal exercise.
Maximal Heart rate | through study completion, an average of 1 year
  the maximum heart rate achieved during intense or maximal exercise.
Maximal Blood pressure | through study completion, an average of 1 year
  the blood pressure in the end of intense or maximal exercise.

SECONDARY OUTCOMES:
Ventilation Anaerobic Threshold | through study completion, an average of 1 year
  Ventilatory Threshold (VT) describes the inflection point for ventilation during an incremental exercise test.

CONTACTS AND LOCATIONS:
Overall Officials: Gur Mainzer, MD, Principal Investigator — The Baruch Padeh Medical Center, Poriya
Locations (1):
- The BARUCH PADEH Medical Center, Poriya, Tiberias, The Lower Galilee, Israel

IPD SHARING:
Plan to Share IPD: No